CLINICAL TRIAL: NCT06210711
Title: Prevention of Posttraumatic Stress: A Randomized Controlled Trial of Brief Prolonged Exposure Therapy for Injured Individuals Admitted to a Level I Trauma Center
Brief Title: Trauma BPE Prolonged Exposure Therapy for Injured Individuals Admitted to a Level I Trauma Center
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Baylor Research Institute (Other)
Collaborators: Froedtert Hospital (Other); Medical College of Wisconsin (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 024-127
Record Dates: First submitted 2024-01-08; First posted 2024-01-18 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Traumatic Injury; PTSD; Posttraumatic Stress Disorder
Keywords: PTSD; Traumatic injury; Posttraumatic stress disorder
MeSH Terms: conditions — Wounds and Injuries; Stress Disorders, Post-Traumatic | interventions — Therapeutics

STUDY DESIGN:
Intervention Model Description: Participants will be allocated 1:1 into the Brief PE intervention or treatment as usual control group.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment as Usual (Placebo Comparator): Participants in the Treatment as Usual group (TAU) will not receive the Brief PE therapy, but the standard clinical treatment received by all patients admitted to BUMC, BSWMC Temple or FH/MCW trauma centers. Treatment as usual participants will have follow-up assessments at 1, 3, and 6 months from Baseline.
  Interventions: Behavioral: Treatment as Usual
- Brief Prolonged Exposure (Experimental): Participants in the experimental group will receive Brief Prolonged Exposure Therapy. In addition to the standard clinical treatment received by all patients at BUMC, BSWMC Temple and FH/MCW (treatment as usual), participants randomized to the intervention condition will also receive three 60-minute sessions of Brief PE. Participants in the BPE group will complete a screener and then questionnaires/interviews at 1, 2, and 6 months from Baseline.
  Interventions: Behavioral: Brief Prolonged Exposure Therapy

INTERVENTIONS:
Behavioral: Treatment as Usual — Standard clinical treatment received by all patients admitted to BUMC, BSWMC Temple or FH/MCW trauma centers. At BUMC and FH/MCW, this may include an evaluation by a licensed psychologist or psychiatrist and continued follow-up psychotherapy and/or medication as needed. At BSWMC Temple this may include an evaluation by a licensed psychiatrist and follow up treatment as needed. In all locations this therapy does not consist of trauma-focused therapy and will be summarized in the analysis as a part of standard of care.
  Arms: Treatment as Usual
Behavioral: Brief Prolonged Exposure Therapy — Brief PE will include 3 therapy sessions, each lasting approximately 60 minutes. The treatment is manualized and has been successfully implemented and evaluated in other challenging environments (i.e., Emergency Department. Trauma center). Brief PE includes education about common reactions to trauma, breathing retraining, prolonged (repeated) imaginal exposure to trauma memories, repeated in vivo/behavioral exposure to situations that participants are avoiding due to trauma-related fear, and discussion of thoughts and feelings related to exposure exercises. This discussion addresses patients' unrealistic beliefs about themselves and the world. In addition, patients are given homework to complete between each session (breathing practice, listening to the session recording, and completing behavioral exposures).
  Arms: Brief Prolonged Exposure

SUMMARY:
The purpose of this research is to determine if a brief treatment method is effective for preventing posttraumatic stress disorder (PTSD) and a number of other concerns following injury.

DETAILED DESCRIPTION:
This is a prospective randomized controlled trial examining the efficacy of brief Prolonged Exposure Therapy (Brief PE) delivered to individuals admitted to a Level I Trauma Center to reduce PTSD symptoms. The overall goal of this project is to test a Brief PE (three 60-minute sessions) to reduce psychological distress after injury and to mitigate long-term post-injury distress including PTSD as well as secondary health outcomes (including depression, general anxiety, pain, and quality of life) at 1, 3, and 6 months from baseline. The intervention group (Brief PE) will be compared to standard clinical care with treatment as usual (TAU).

ELIGIBILITY:
Inclusion Criteria:

* Between the ages of 18 and 75 years old.
* Admitted to Baylor University Medical Center at Dallas (BUMC), Baylor Scott & White Medical Center at Temple (BSWMC), or Froedtert Hospital and the Medical College of Wisconsin (FH/MCW) Level 1 Trauma Center

Exclusion Criteria:

* Patients in police custody
* Patients not fluent in English
* Patients with severe cognitive impairment
* Patients who are acutely suicidal
* Patients with active psychosis

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2024-02-28 (Actual); Primary Completion 2027-03 (Estimated); Study Completion 2027-09 (Estimated)

PRIMARY OUTCOMES:
Clinician Administered PTSD Scale for DSM-5 (CAPS-5) | Baseline, 1-month, 3-month, 6-months
  The CAPS-5 is a 30-item, structured interview that assesses PTSD symptoms and makes a diagnostic determination based on the DSM-5 criteria and is considered the gold standard of PTSD assessment. Questions assess for PTSD symptoms corresponding to the 4 DSM-5 clusters of re-experiencing, avoidance, changes in mood and cognition, and arousal and hyperactivity, and includes questions on duration, impact of symptoms, distress and impact of symptoms on social and occupational functioning. The interviewer rates participant responses to symptom questions on a 5-point scale of frequency and severity, from 0 ("Absent") to 4 ("Extreme/incapacitating").
PTSD Checklist for DSM-5 (PCL-5) | Baseline, 1-month, 3-month, 6-months
  The PCL-5 is a 20-item, self-report measure that assesses history of traumas and PTSD symptom severity over the last month according to the DSM-5 criteria.

SECONDARY OUTCOMES:
Patient Health Questionnaire (PHQ-9) | Baseline, 1-month, 3-month, 6-months
  The PHQ-9 is a brief self-report measure of major depressive disorder. The PHQ-9 is a valid measure of depression for population-based studies and clinical populations with a cut off score of equal to or greater than 10 as the diagnostic for current depression.
The Generalized Anxiety Disorder 7-Item (GAD-7) | Baseline, 1-month, 3-month, 6-months
  The GAD-7 is a 7-item questionnaire that measures severity of anxiety. Response options are "not at all," "several days," "more than half the days," and "nearly every day," scored as 0, 1, 2, and 3, respectively. Therefore, GAD-7 scores range from 0 to 21, with scores of 5, 10, and 15 representing mild, moderate, and severe anxiety symptom levels, respectively.
Brief Pain Inventory-Short Form (BPI-SF) | Baseline, 1-month, 3-month, 6-months
  The BPI-SF has 9 items that measure the severity and impact of pain on daily function, with scores ranging from 0 (no pain and no interference) to 10 (pain as bad as one can imagine and complete interference) over the past 24 hours.
Quality of Life Enjoyment and Satisfaction Questionnaire-Short Form (Q-LES-Q-SF) | 1-month, 3-month, 6-months
  Th3 Q-LES-Q-SF examines life satisfaction over the past week. The 16 items are rated on a 5-point scale from 1 "very poor" to 5 "very good" with scores from items added together and reported as a maximum possible score in percentage.

CONTACTS AND LOCATIONS:
Overall Officials: Ann Marie Warren, PhD, Principal Investigator — Baylor Scott & White Research Institute
Locations (3):
- United States (3):
  - Baylor University Medical Center, Dallas, Texas
  - Baylor Scott & White Medical Center - Temple, Temple, Texas
  - Froedtert & Medical College of Wisconsin, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: Yes
Data from this study will be submitted to the National Institute of Mental Health (NIMH) Data Archive (NDA) at the National Institutes of Health (NIH). The NDA is a large database where de-identified study data from many NIH studies are stored and managed. Sharing your de-identified study data helps researchers learn new and important things about brain science more quickly than before. The following data will be submitted: Age, DSM-5 crosscutting assessment, PHQ-9, and the GAD-7.